CLINICAL TRIAL: NCT00779584
Title: A Phase 1 Dose-Escalation Study of SCH 900776 as Monotherapy and in Combination With Gemcitabine in Subjects With Advanced Solid Tumors or Lymphoma
Brief Title: A Dose-escalation Study of MK-8776 (SCH 900776) With and Without Gemcitabine in Participants With Solid Tumors or Lymphoma (MK-8776-002/P05248)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05248; MK-8776-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms | interventions — MK-8776; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 (Experimental): Participants received MK-8776 10 mg/m^2 given as monotherapy as an intravenous (IV) infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 800 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine
- MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 (Experimental): Participants received MK-8776 20 mg/m^2 given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 800 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine
- MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 (Experimental): Participants received MK-8776 40 mg/m^2 given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 800 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine
- MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 (Experimental): Participants received MK-8776 80 mg/m^2 given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 800 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine
- MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 (Experimental): Participants received MK-8776 112 mg/m^2 given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 800 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine
- MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 (Experimental): Participants received MK-8776 80 mg/m^2 given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 1000 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine
- MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 (Experimental): Participants received MK-8776 112 mg/m^2 given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 1000 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine
- MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 (Experimental): Participants received MK-8776 150 mg/m^2 given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 1000 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine
- MK-8776 200mg+Gemcitabine 1000mg/m^2 (Experimental): Participants received MK-8776 200 mg given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 1000 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
  Interventions: Drug: MK-8776; Drug: Gemcitabine

INTERVENTIONS:
Drug: MK-8776 — IV infusion
  Other Names: SCH 900776
Drug: Gemcitabine — IV infusion
  Other Names: GEMZAR®

SUMMARY:
This study of MK-8776 (SCH 900776) will evaluate its safety and tolerability when given as monotherapy or in combination with gemcitabine to participants with advanced solid tumors or lymphoma. Participants will be enrolled in cohorts that will receive sequentially higher doses of MK-8776 in combination with standard doses of gemcitabine The recommended combination doses for a Phase 2 trial (combination-RP2D) will be determined based on safety and biological activity. Up to 10 to 15 additional participants may be studied at the combination-RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of an advanced solid tumor malignancy or lymphoma (non-Hodgkin's or Hodgkin's lymphoma).
* Must have histological or cytological evidence of malignancy.
* Must have an advanced malignancy, metastatic or unresectable. For Part A of the study, the metastatic or unresectable malignancy should have recurred or progressed following standard therapy or failed standard therapy; or for which no standard therapy currently exists, or for which they are not candidates for standard therapy. For Parts B and C of the study, participants with advanced tumors for which gemcitabine is considered standard therapy (eg, pancreatic cancer), may be enrolled without having received prior gemcitabine. Standard therapy is defined as therapy that is approved in a particular line of therapy or considered as standard of care based on published peer reviewed data in a specific line of therapy.
* Gemcitabine-naïve participants with tumors known to be responsive to gemcitabine or participants previously treated with gemcitabine who did not progress while on treatment or who are currently still responding to treatment should only be enrolled in cohorts for which gemcitabine doses are >=1000 mg/m². Participants previously treated with gemcitabine, whose disease has progressed wile on treatment, can be enrolled to any part.
* Must be ambulatory with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants (and/or parent/guardian for participants who otherwise are unable to provide independent consent) must be willing to give written informed consent and able to adhere to dose and visit schedules.
* Female participants of childbearing potential must have a negative pregnancy test within 7 days of first dose of protocol therapy.
* Female participants of childbearing potential and male participants whose sexual partners are of childbearing potential must agree to abstain from sexual intercourse or to use an acceptable method of contraception during the study and for 90 days following the last dose of protocol therapy. Acceptable methods of contraception include condoms (male or female) with or without spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device (IUD), oral or injectable hormonal contraceptive, and surgical sterilization (eg, hysterectomy or tubal ligation).
* Must have adequate bone marrow reserve as evidenced by a white blood cell (WBC) count >=3,000/ μL, absolute neutrophil count (ANC) >=1,500/μL AND platelet count >=100,000/μL.
* Must have adequate renal function as evidenced by a serum creatinine level <=1.5 x upper limit of normal (ULN) or a calculated creatinine clearance >60 mL/min.
* Participants, except those with known Gilbert's Syndrome, must have adequate hepatic function as evidenced by a serum bilirubin level <=1.5 x the ULN AND serum levels of aspartate and alanine aminotransferase (AST/ALT) levels <=3 x the ULN for the reference lab (participants with known hepatic metastases must have serum AST/ALT levels <=5 x the ULN for the reference lab).
* Must be recovered from the effects of any prior surgery, radiotherapy or systemic antineoplastic therapy.

Exclusion Criteria:

* Has a known hypersensitivity to MK-8776 or gemcitabine or to any of their excipients or has received therapy with another Checkpoint kinase 1 (CHK1) inhibitor.
* Has received any prohibited medication more recently than the indicated washout period prior to first dose of protocol therapy or must continue to receive prohibited medications. Prohibited medications: cytochrome P450 1A2 inhibitors, any chemotherapy, or investigational drugs.
* Has significant underlying cardiac conduction system abnormalities such as bifascicular or greater block (eg, right bundle branch block with left anterior hemiblock or first degree atrioventricular block), fixed-rate pacemaker, or chronic atrial fibrillation with variable ventricular rate.
* Has persistent, unresolved Common Terminology Criteria for Adverse Events (CTCAE) v 3.0 >=Grade 2 drug-related toxicity (except alopecia, erectile impotence, hot flashes, and decreased libido) associated with previous treatment.
* Has known human immunodeficiency virus (HIV), hepatitis B, hepatitis C, or a known history of liver cirrhosis or active alcohol abuse.
* Is New York Heart Association (NYHA) Class III.
* Has any other medical or psychiatric condition that, in the opinion of the investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.
* Has undergone major surgery within 3 weeks prior to first study drug administration after enrollment.
* Has central nervous system (CNS) or leptomeningeal metastases.
* Has received radiation therapy within 3 weeks prior to first study drug administration after enrollment or radiation therapy to >25% of bone marrow.
* Has received >3 prior chemotherapy regimens (may have received prior gemcitabine). A participant may not have experienced any CTCAE v 3.0 >Grade 1 myelotoxicity (neutropenia and/or thrombocytopenia) with any prior regimen, including gemcitabine. Participants with >3 prior chemotherapy regimens, one or more of which were targeted, nonmyelosuppressive agents, may be considered on a case-by-case basis after discussion with the sponsor.
* Has undergone previous allogeneic or autologous stem cell transplant.
* Has had any of the following within 6 months prior to first study drug administration after enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or seizure disorder.
* Has a known bleeding diathesis, eg, hemophilia.
* Has a baseline QTc interval >450 msec (ie, CTCAE v 3.0 Grade ≥2) at screening (within 21 days prior to 1st dose of MK-8776, mean of triplicate readings within approximately 5 minutes).
* History of risk factors for Torsades de Pointes, including clinical history of heart failure, hypo- or hyperkalemia or hypomagnesemia (supplementation or other appropriate interventions to bring levels within normal institutional limits prior to administration of MK-8776 is acceptable), or family history of Long QT Syndrome.
* Currently a smoker and/or is likely to smoke during the study.
* Female participant who is breast-feeding, pregnant, or intends to become pregnant.
* Participating in any other interventional clinical study. (Participants participating in another noninterventional study may be considered after discussion with the sponsor.)
* Part of the staff personnel directly related to this study.
* Family member of one of the investigational staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-10-17 (Actual); Primary Completion 2011-05-28 (Actual); Study Completion 2011-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Daud AI, Ashworth MT, Strosberg J, Goldman JW, Mendelson D, Springett G, Venook AP, Loechner S, Rosen LS, Shanahan F, Parry D, Shumway S, Grabowsky JA, Freshwater T, Sorge C, Kang SP, Isaacs R, Munster PN. Phase I dose-escalation trial of checkpoint kinase 1 inhibitor MK-8776 as monotherapy and in combination with gemcitabine in patients with advanced solid tumors. J Clin Oncol. 2015 Mar 20;33(9):1060-6. doi: 10.1200/JCO.2014.57.5027. Epub 2015 Jan 20. PMID 25605849

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-8776 200mg+Gemcitabine 1000mg/m^2: Participants received MK-8776 200 mg given as a flat dose monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 1000 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
Period: Overall Study
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2
Started | 3 | 3 | 7 | 6 | 7 | 6 | 8 | 3 | 2
Treated | 3 | 3 | 7 | 6 | 7 | 4 | 8 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 7 | 6 | 7 | 6 | 8 | 3 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progression of Disease | 0 | 1 | 2 | 6 | 5 | 1 | 4 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Symptomatic Deterioration | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Ongoing in Study | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-8776 10mg/m^2+Gemcitabine 800mg/m^2: Participants received MK-8776 10 mg/m^2 given as monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 800 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
- Total: Total of all reporting groups
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 7 | 6 | 8 | 3 | 2 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (16.0) | 54.3 (8.6) | 64.0 (16.1) | 55.5 (5.0) | 51.1 (5.7) | 59.0 (13.4) | 59.9 (9.1) | 69.3 (5.5) | 69.0 (8.5) | 58.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 2 | 4 | 2 | 3 | 1 | 2 | 18
  Male | 1 | 3 | 5 | 4 | 3 | 4 | 5 | 2 | 0 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT) During Cycle 0 and Cycle 1 Based on National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE v 3.0)
Description: During Cycle 0, a DLT was defined as: CTCAE v 3.0 Grade 3 neutropenia or thrombocytopenia lasting ≥3 days; any CTCAE v 3.0 Grade 4 neutropenia or thrombocytopenia; neutropenic fever; any CTCAE v. 3.0 ≥ Grade 3 QT interval corrected by Fridericia (QTcF) prolongation of any duration; any other CTCAE v 3.0 Grade 3 or higher nonhematologic toxicity; or Grade 3 elevation of transaminases that resolved prior to administration of next dose(s) of study drug(s); delay in Cycle 1 Day 1 beyond 3 weeks due to continuing toxicity. During Cycle 1, a DLT was defined as: CTCAE v 3.0 Grade 4 neutropenia that persists for ≥7 days; neutropenic fever; CTCAE v 3.0 Grade 4 thrombocytopenia; CTCAE v 3.0 ≥ Grade 3 thrombocytopenia with bleeding; any CTCAE v 3.0 QTc ≥ Grade 3 QTcF prolongation of any duration; any other CTCAE v 3.0 Grade 3 or higher nonhematologic toxicity; or Grade 3 elevation of transaminases that resolved prior to administration of next dose(s) of study drug(s).
Time Frame: Through Cycle 0 and Cycle 1 (Up to 42 days)
Population: The population consisted of all participants who were evaluable for DLT assessment (i.e., completed Cycle 0 and Cycle 1).
Measure: Number; unit: Participants
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 7 | 4 | 6 | 3 | 2
Participants | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could have been any unfavorable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to study treatment. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 72 weeks (Up to approximately 6 weeks after last dose of study treatment)
Population: The population consisted of all participants who received at least one dose of MK-8776.
Measure: Number; unit: Participants
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 7 | 4 | 8 | 3 | 2
Participants | 3 | 3 | 7 | 6 | 7 | 4 | 8 | 3 | 2

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could have been any unfavorable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to study treatment. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximatey 66 weeks
Population: The population consisted of all participants who received at least one dose of MK-8776.
Measure: Number; unit: Participants
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 7 | 4 | 8 | 3 | 2
Participants | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 1

4. Secondary Outcome: MK-8776 Maximum Plasma Concentration (Cmax)
Description: The Cmax of MK-8776 was assessed in Cycle 0 and in Cycle 1. On Day 1 of Cycle 0 and Cycle 1, plasma samples were obtained from all participants before infusion, at end of infusion of MK-8776 (Cycle 0) or gemcitabine (Cycle 1), and at 0.25, 1, 3, 6, 8, 24 and 48 hours after completion of MK-8776 infusion.
Time Frame: At end of infusion of MK-8776 (Cycle 0) or gemcitabine (Cycle 1), and at 0.25, 1, 3, 6, 8, 24 and 48 hours after completion of MK-8776 infusion
Population: The population consisted of all participants who received at least two cycles of study treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 7 | 4 | 8 | 3 | 2
ng/mL
  Cycle 0 (n=3, 3, 7, 6, 7, 4, 8, 3, 2) | 414 (257) | 1010 (197) | 1220 (366) | 4970 (1500) | 5270 (3730) | 2960 (1290) | 6210 (2160) | 6220 (2550) | 4860 (NA) — By Sponsor convention, standard deviations are only calculated when the number of participants analyzed (n) ≥ 3.
  Cycle 1 (n=3, 3, 7, 5, 6, 4, 6, 1, 2) | 445 (249) | 1650 (1520) | 962 (454) | 3700 (1930) | 4710 (2310) | 3610 (2290) | 4690 (2610) | 4940 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3. | 3700 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3.

5. Secondary Outcome: MK-8776 Area Under the Curve of the Plasma Concentration Versus Time From Time Zero to the Time of the Last Analytically Quantifiable Concentration (AUC0-last)
Description: AUC0-last was assessed in Cycle 0 and in Cycle 1. On Day 1 of Cycle 0 and Cycle 1, plasma samples were obtained from all participants before infusion, at end of infusion of MK-8776 (Cycle 0) or gemcitabine (Cycle 1), and at 0.25, 1, 3, 6, 8, 24 and 48 hours after completion of MK-8776 infusion. AUC0-last was calculated by the linear trapezoidal method.
Time Frame: as for outcome 4
Population: The population consisted of all participants who received at least two cycles of study treatment.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 7 | 4 | 8 | 3 | 2
ng*hr/mL
  Cycle 0 (n=3, 3, 7, 6, 7, 4, 8, 3, 2) | 565 (171) | 1400 (448) | 2250 (948) | 5060 (1920) | 9050 (5500) | 4040 (1010) | 9240 (5740) | 18500 (8000) | 8440 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3.
  Cycle 1 (n=3, 3, 7, 5, 6, 4, 6, 1, 2) | 539 (307) | 1570 (423) | 1900 (859) | 4540 (1660) | 10300 (6370) | 4660 (815) | 6900 (3120) | 13000 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3. | 16900 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3.

6. Secondary Outcome: Time of MK-8776 Cmax (Tmax)
Description: The time of Cmax of MK-8776 was assessed in Cycle 0 and in Cycle 1. On Day 1 of Cycle 0 and Cycle 1, plasma samples were obtained from all participants before infusion, at end of infusion of MK-8776 (Cycle 0) or gemcitabine (Cycle 1), and at 0.25, 1, 3, 6, 8, 24 and 48 hours after completion of MK-8776 infusion.
Time Frame: as for outcome 4
Population: The population consisted of all participants who received at least two cycles of study treatment.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 7 | 4 | 8 | 3 | 2
hr
  Cycle 0 (n=3, 3, 7, 6, 7, 4, 8, 3, 2) | 0.27 (0.03) | 0.26 (0.01) | 0.29 (0.06) | 0.24 (0.03) | 0.30 (0.08) | 0.26 (0.05) | 0.23 (0.02) | 0.48 (0.02) | 0.49 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3.
  Cycle 1 (n=3, 3, 7, 5, 6, 4, 6, 1, 2) | 0.26 (0.01) | 0.27 (0.02) | 0.35 (0.13) | 0.25 (0.06) | 0.28 (0.06) | 0.26 (0.03) | 0.23 (0.01) | 0.50 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3. | 0.57 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3.

7. Secondary Outcome: MK-8776 Terminal Phase Half-Life (t1/2)
Description: The t1/2 of MK-8776 was assessed in Cycle 0 and in Cycle 1. On Day 1 of Cycle 0 and Cycle 1, plasma samples were obtained from all participants before infusion, at end of infusion of MK-8776 (Cycle 0) or gemcitabine (Cycle 1), and at 0.25, 1, 3, 6, 8, 24 and 48 hours after completion of MK-8776 infusion.
Time Frame: as for outcome 4
Population: The population consisted of all participants who received at least two cycles of study treatment.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg+Gemcitabine 1000mg/m^2
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 7 | 4 | 8 | 3 | 3
hr
  Cycle 0 (n=3, 3, 7, 6, 7, 4, 8, 3, 2) | 6.29 (1.97) | 9.33 (5.09) | 8.45 (2.95) | 7.44 (0.435) | 5.94 (1.62) | 8.13 (1.30) | 7.14 (1.90) | 9.46 (2.11) | 6.30 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3.
  Cycle 1 (n=3, 3, 6, 6, 7, 4, 7, 1, 2) | 6.24 (2.03) | 8.57 (4.54) | 8.23 (1.71) | 9.01 (2.51) | 7.29 (1.26) | 7.87 (2.11) | 7.98 (1.21) | 7.59 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3. | 9.89 (NA) — By Sponsor convention, standard deviations are only calculated when n ≥ 3.

ADVERSE EVENTS:
Time Frame: Up to approximately 72 weeks (Up to approximately 6 weeks after last dose of study treatment)
Description: The population consisted of all participants who received at least one dose of MK-8776.
Groups:
- MK-8776 200mg Flat Dose+Gemcitabine 1000mg/m^2: Participants received MK-8776 200 mg given as a flat dose monotherapy as an IV infusion on Cycle 0 Day 1 and as combination therapy with gemcitabine 1000 mg/m^2 starting with Cycle 1 on Days 1 and 8 of a 21-day treatment cycle.
Arm/Group | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 | MK-8776 200mg Flat Dose+Gemcitabine 1000mg/m^2
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 3/7 | 1/6 | 2/7 | 3/4 | 4/8 | 0/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 6/6 | 7/7 | 4/4 | 8/8 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 (N=3) | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 (N=3) | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 (N=7) | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 (N=6) | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 (N=7) | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 (N=4) | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 (N=8) | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 (N=3) | MK-8776 200mg Flat Dose+Gemcitabine 1000mg/m^2 (N=2)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MASTOIDITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8776 10mg/m^2+Gemcitabine 800mg/m^2 (N=3) | MK-8776 20mg/m^2+Gemcitabine 800mg/m^2 (N=3) | MK-8776 40mg/m^2+Gemcitabine 800mg/m^2 (N=7) | MK-8776 80mg/m^2+Gemcitabine 800mg/m^2 (N=6) | MK-8776 112mg/m^2+Gemcitabine 800mg/m^2 (N=7) | MK-8776 80mg/m^2+Gemcitabine 1000mg/m^2 (N=4) | MK-8776 112mg/m^2+Gemcitabine 1000mg/m^2 (N=8) | MK-8776 150mg/m^2+Gemcitabine 1000mg/m^2 (N=3) | MK-8776 200mg Flat Dose+Gemcitabine 1000mg/m^2 (N=2)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 2 (7) | 4 (13) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (4) | 3 (6) | 1 (1) | 4 (6) | 1 (2) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EUSTACHIAN TUBE OBSTRUCTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIDDLE EAR EFFUSION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (5) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
DENTAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
GINGIVAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (5) | 1 (1) | 2 (5) | 3 (3) | 4 (6) | 3 (5) | 2 (3) | 3 (3) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SALIVARY GLAND ENLARGEMENT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (3) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATHETER SITE PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
EARLY SATIETY (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 2 (4) | 5 (6) | 5 (7) | 6 (9) | 4 (10) | 4 (6) | 1 (1) | 0 (0)
GENERALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION SITE PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (2) | 1 (2) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BILIARY DILATATION (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATIC PAIN (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 1 (1)
CANDIDIASIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TINEA MANUUM (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BREATH SOUNDS ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (25) | 1 (5) | 2 (7) | 3 (5) | 1 (3)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (4) | 3 (4) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (8) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPOGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOSMIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEDATION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLAT AFFECT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLADDER PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHROMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RALES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN TIGHTNESS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.